CLINICAL TRIAL: NCT06068530
Title: A Cluster-randomised, Open-label Trial to Compare the Impact of Combined Mass Vaccine and Drug Administrations, Mass Drug Administration, Mass Vaccinations, or no Intervention on Plasmodium Falciparum Malaria Transmission
Brief Title: Mass Vaccine and Drug Administration, Bangladesh
Acronym: MVDA
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MAL23002
Record Dates: First submitted 2023-08-22; First posted 2023-10-05 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-02

CONDITIONS: Plasmodium Falciparum Malaria
Keywords: Plasmodium Falciparum Malaria; Malaria Vaccine; Malaria Drug Administrations
MeSH Terms: conditions — Malaria, Falciparum

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- MDA + Vaccine (Active Comparator): The participants in MVDA villages will receive R21/Matrix M at M0, M1, M2, and a booster M12 plus DHA/piperaquine and a SLD-PQ at M0, M1, and M2
  Interventions: Drug: DHA/piperaquine and a SLD-PQ; Biological: Study vaccine R21/Matrix-M™
- MDA only (Active Comparator): The participants in MDA only villages will receive DHA/piperaquine and a SLD-PQ at M0, M1, and M2
  Interventions: Drug: DHA/piperaquine and a SLD-PQ
- Vaccine only (Active Comparator): The participants in vaccine only villages will receive R21/Matrix M at M0, M1, M2, and a booster M12
  Interventions: Biological: Study vaccine R21/Matrix-M™
- Control (No Intervention): The participants in control will receive MVDA at the end of the 24th month assuming that MVDA is found to be safe and effective. During M0 to M24, the comparison villages will receive the standard of care as per national malaria treatment guidelines.

INTERVENTIONS:
Drug: DHA/piperaquine and a SLD-PQ — Participants in Arms 1 and 2 will receive three rounds of antimalarial drugs - each round starting on the day of vaccination (Day 0) at Study Months 0, 1, and 2. Each round consists of three daily doses of co-formulated dihydroartemisinin/piperaquine on Day 0, 1, and 2 (i.e. the day of vaccination and each day for 2 days after). The drug dose is based on the weight of the participant at the first visit (M0D0). Dihydroartemisinin/piperaquine tablets (Shanghai Fosun Pharmaceutical Co., Ltd.) for adult participants each contain 40 mg dihydroartemisinin and 320 mg piperaquine with a therapeutic dose range between 2-10 mg/kg/day dihydroartemisinin and 16-26 mg/kg/dose piperaquine. In addition, each participant will receive a single low dose primaquine on the day of vaccination (Day 0; Table 4). One single low dose primaquine of approximately 0.25 mg/kg (Thai Government Pharmaceutical Organisation) will be administered. Children under 10kg do not receive PQ.
  Arms: MDA + Vaccine; MDA only
Biological: Study vaccine R21/Matrix-M™ — The mixing prior to administration strategy will involve withdrawal of 0.5 mL antigen from one vial of R21 Malaria vaccine and adding it to Matrix-M1 vial. 0.5 mL of R21 antigen shall be withdrawn from another vial of R21 Malaria vaccine and be added to the same Matrix-M1 vial. The total volume in Matrix-M1 vial will be 1.5 mL. After addition the content will be mixed gently, and 0.75 mL of the mixture will be withdrawn and administered to participants. Each dose of 0.75mL (after mixing of R21 with Matrix-M1) will contain 10 µg of R21 and 50 µg for participants 14 years and older. In children up to 14 years a 5 μg will be used.
  Arms: MDA + Vaccine; Vaccine only

SUMMARY:
This is an open i.e. not blinded, cluster-randomised, controlled intervention study. The study will use a factorial design to estimate the protective effectiveness of mass drug administrations, mass vaccinations, combined mass vaccinations and drug administrations versus the current standard of care.

DETAILED DESCRIPTION:
Trial Activities: The investigators are most interested in the combined effect of mass administration of vaccines and drugs on malaria transmission. Can Mass Vaccine and Drug Administrations (MVDA) reduce the parasite prevalence in intervention villages compared to control villages which did not receive the intervention? The entire village population will be enrolled at study start and followed for two years after D0, the first day of the interventions in the intervention villages. The village population is a dynamic cohort with new members entering the cohort by birth or immigration and other members leaving the cohort due to emigration or death. Newcomers entering villages will receive MVDA as soon as feasible and as appropriate (dependent on age). Secondly, the investigators want to know how effective the individual components of the intervention, mass vaccinations and mass drug administrations are in relation to MVDA?

Hanako Foundation funded this study. Grant reference number: B9R05700

ELIGIBILITY:
Inclusion Criteria:

* Current residence in a study village irrespective of permanence
* Age 6 months and above (no upper age limit)
* Written informed consent provided by participants (or a parent/guardian in case the participant is under 18 years old)

Exclusion Criteria:

* Pregnancy, plan to get pregnant, or breastfeeding.
* Acute illness requiring intervention
* A history of an adverse reaction to study drugs/vaccine and prior receipt of any other malaria vaccine or enrolment in another intervention trial.

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10000 (Estimated)
Dates: Start 2025-02-15 (Actual); Primary Completion 2028-02-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Falciparum malaria incidence by study groups | Data will be collected for two years following baseline intervention (Month 0 to Month 24)
  Falciparum malaria incidence will be determined by the number of clinical falciparum malaria cases confirmed by Rapid diagnostic test (RDT) or microscopy to determine the overall protective efficacy against clinical falciparum malaria among study groups.
  The investigators will look for the presence of axillary temperature ≥37.5°C AND P. falciparum positive RDT or microscopy as a primary case definition of clinical falciparum malaria.
Falciparum malaria prevalence by study groups | PCR for malaria detection from DBS will be collected at 6th month intervals until two years following baseline intervention (Month 0, Month 6, Month 12, Month 18 and Month 24)
  Falciparum malaria prevalence will be determined by the number of positive falciparum confirmed by dried blood spots (DBS) polymerase chain reaction (PCR) malaria detection method during cross-sectional surveys to determine the overall protective efficacy against subclinical P. falciparum among study groups.
  * The investigators will collect dried blood spots to detect malaria during cross-sectional surveys from the healthy participants.
  * Those who have axillary temperature ≥37.5°C AND P. falciparum positive RDT or microscopy will receive treatment according to national treatment guidelines.
Overall percentage of falciparum malaria positivity by study groups | DBS: Month 0, Month 6, Month 12, Month 18 and Month 24 and Clinical malaria data for two year following intervention
  The percentage of falciparum malaria positivity will be determined by the number of falciparum positives detected by PCR, RDT or microscopy to determine overall protective efficacy against clinical and subclinical falciparum malaria among study groups. Dried blood spots to detect malaria from by PCR will be collected at baseline and every six months until two years. Clinical malaria data detected by rapid diagnostic test or microscopy will be collected for two years following intervention.
  * The investigators will look for the presence of axillary temperature ≥37.5°C AND P. falciparum positive RDT or microscopy as a primary case definition of clinical malaria.
  * The investigators will collect dried blood spots to detect malaria during cross-sectional surveys from the healthy participants.

SECONDARY OUTCOMES:
The incidence of Deaths related to falciparum malaria among study groups | Data will be collected for two years following baseline intervention (Month 0 to Month 24)
  The number of Deaths related to falciparum malaria (confirmed by RDT or microscopy) will be recorded for two year following intervention. Death rate among study groups will be compared
The incidence of severe malaria disease among study groups | Data will be collected for two years following baseline intervention (Month 0 to Month 24)
  The number of Severe malaria diseases (according to WHO criteria) will be recorded for two years following intervention and the incidences will be compared among study groups.
  Primary case definition of severe malaria:
  * Presence of P. falciparum (RDT positive or microscopy positive); AND one of more of the following criteria of disease severity:
  * Prostration
  * Respiratory distress
  * Blantyre coma score ≤ 3
  * Seizures: 2 or more
  * Hypoglycemia < 2.2 mmol/L
  * Acidosis BE ≤-8.0 mmol/L
  * Lactate ≥ 5.0 mmol/L
  * Anemia < 5.0 g/dL
  * Acute kidney injury
  * Pulmonary oedema
  * Significant bleeding
  * Shock (systolic BP <70mm Hg); AND Without any of the following criteria of co- morbidity
  * Pneumonia (confirmed by X-ray)
  * Meningitis (confirmed by CSF examination)
  * Sepsis (with Positive blood culture)
  * Gastroenteritis with dehydration
The incidence of severe anaemia among study groups | Data will be collected for two years following baseline intervention (Month 0 to Month 24)
  The number of severe anemia cases will be recorded for two years following interventions among all participants and the proportions will be compared among study groups Severe anaemia due to severe malaria according to WHO criteria
  * Anaemia < 5.0 g/dL
  * Requires blood transfusion according to National guidelines
Vivax malaria incidence by study groups | Data will be collected for two years following baseline intervention (Month 0 to Month 24)
  Vivax malaria incidence will be determined by the number of clinical vivax malaria cases confirmed by RDT or microscopy to determine the overall protective efficacy against clinical vivax malaria among study groups.
  The investigators will look for the presence of axillary temperature ≥37.5°C AND P.vivax positive RDT or microscopy as a primary case definition of clinical vivax malaria.
Vivax malaria prevalence by study groups | PCR for malaria detection from DBS will be collected at 6th month intervals until two years following baseline intervention (Month 0, Month 6, Month 12, Month 18 and Month 24)
  Vivax malaria prevalence will be determined by the number of positive vivax confirmed by dried blood spots PCR malaria detection method during cross-sectional surveys to determine the overall protective efficacy against subclinical P. vivax among study groups.
  * The investigators will collect dried blood spots to detect malaria during cross-sectional surveys from the healthy participants.
  * Those who have axillary temperature ≥37.5°C AND P. vivax positive RDT or microscopy will receive treatment according to national treatment guideline.
Overall percentage of vivax malaria positivity by study groups | DBS: Month 0, Month 6, Month 12, Month 18 and Month 24 and Clinical malaria data for two year following intervention
  The percentage of vivax malaria positivity will be determined by the number of vivax positives detected by PCR, RDT or microscopy to determine overall protective efficacy against clinical and subclinical vivax malaria among study groups. Dried blood spots to detect malaria from by PCR will be collected at baseline and every six months until two years. Clinical malaria data detected by rapid diagnostic test or microscopy will be collected for two years following intervention.
  * The investigators will look for the presence of axillary temperature ≥37.5°C AND P. vivax positive RDT or microscopy as a primary case definition of clinical malaria.
  * The investigators will collect dried blood spots to detect malaria during cross-sectional surveys from the healthy participants.
The incidence of adverse events | All adverse events which occur after administration of the first dose of the study drugs until one month after last dose of drugs or vaccine will be recorded. This data will be collected from Month 0 to month 24.
  The number of events will be assessed and graded according to Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 among all participants and compared among study groups to determine the safety and reactogenicity
  * Occurrence of solicited local and/or systemic reactogenicity signs and symptoms for 7 days following the intervention ((a) R21 adjuvanted with Matrix-M b) mass drug administration with DHA/piperaquine plus SLDPQ c) vaccine and MDA combined)
  * Occurrence of unsolicited adverse events for 28 days following the intervention
  * Occurrence of serious adverse events for the duration of the trial
The concentration of antibodies against Plasmodium falciparum circumsporozoite (anti-NANP total IgG antibody) among subset of randomly selected participants from vaccinated and no intervention group. | One month after the completion of the third dose (at Study month 3), and one month after the booster dose (at Study Month 13)
  * Comparison of immunogenicity (antibody responses to CSP) in the R21/MM vaccination group with those in the a) combined group vaccine plus MDA b) control group (mass drug administration with DHA/piperaquine plus SLDPQ)
  * ELISA to quantify antibodies to the vaccine components (regions of the CS antigen including the NANP repeat region and other elements of the protein as well as anti HBs)
Prevalence of molecular markers for drug resistant P. falciparum | Data will be collected for two years following baseline intervention (Month 0 to Month 24)
  The presence (Number) of molecular markers for drug resistant P. falciparum such as Kelch 13 mutations, plasmepsin 2 and mdr1 will be measured from DBS samples for all falciparum positive cases to determine the prevalence among test participants in each study group.
The acceptability of the intervention will be assessed by coverage (The number of residents participating in the interventions) reported as percentage of the target population participating in the intervention. | Month 3 and Month 13
The acceptability of the intervention will be assessed by mixed social science methods, in depth interviews and Focus group discussions. | Data will be collected for two years following baseline intervention (Month 0 to Month 24)
The incidence of clinical falciparum malaria confirmed by RDT or microscopy among vaccinated and drug administered participants in compare to unvaccinated and no drug-administered participants living in standard-of-care villages. | Data will be collected for two years following baseline intervention (Month 0 to Month 24)
  To determine the direct protective efficacy of the combined intervention MVDA against falciparum malaria infection. Data on falciparum malaria infection confirmed by RDT or microscopy will be collected and measured.
The incidence of clinical falciparum malaria confirmed by RDT or microscopy among vaccinated participants in compare to unvaccinated participants living in standard-of-care villages. | Data will be collected for two years following baseline intervention (Month 0 to Month 24)
  To determine direct protective efficacy of the vaccination alone against falciparum malaria infection. Data on falciparum malaria infection confirmed by RDT or microscopy will be collected to measure incidence.
The incidence of clinical falciparum malaria confirmed by RDT or microscopy among drug administered participants in compare to no drug-administered participants living in standard-of-care villages. | Data will be collected for two years following baseline intervention (Month 0 to Month 24)
  To determine direct protective efficacy of the mass drug administration alone against falciparum malaria infection. Data on falciparum malaria infection confirmed by RDT or microscopy will be collected to measure incidence.
The incidence of clinical falciparum malaria confirmed by RDT or microscopy among unvaccinated and no drug-administered people living in intervention clusters relative to unvaccinated and no drug-administered people living in standard-of-care villages. | Data will be collected for two years following baseline intervention (Month 0 to Month 24)
  To determine indirect protective efficacy of the combined intervention MVDA observed against falciparum malaria infection. Data on falciparum malaria infection confirmed by RDT or microscopy will be collected and measured.
The incidence of clinical falciparum malaria confirmed by RDT or microscopy among unvaccinated people living in intervention clusters relative to unvaccinated people living in standard-of-care villages. | Data will be collected for two years following baseline intervention (Month 0 to Month 24)
  To determine Indirect protective efficacy of the vaccination alone observed against falciparum malaria infection. Data on falciparum malaria infection confirmed by RDT or microscopy will be collected and measured.
The incidence of clinical falciparum malaria confirmed by RDT or microscopy among no drug-administered people living in intervention clusters relative to no drug-administered people living in standard-of-care villages. | Data will be collected for two years following baseline intervention (Month 0 to Month 24)
  To determine indirect protective efficacy of the mass drug administration alone observed against falciparum malaria infection. Data on falciparum malaria infection confirmed by RDT or microscopy will be collected and measured.

CONTACTS AND LOCATIONS:
Overall Officials: Lorenz von Seidlein, Principal Investigator — Mahidol University
Locations (2):
- Bangladesh (2):
  - Alikadam Upazila Health Complex, Bāndarban
  - Lama Upazila Health Complex, Lāma

IPD SHARING:
Plan to Share IPD: Yes
With participant's consent, participant's data and results from blood analyses stored in the database may be shared according to the terms defined in the MORU data sharing policy with data repositories such as the WorldWide Antimalarial Resistance Network (WWARN, terms of submission here: http://www.wwarn.org/tools-resources/terms-submission) or other researchers to use in the future. All personal information will be anonymised so that no individual can be identified from their treatment records, through interviews, or from mapping data.